CLINICAL TRIAL: NCT03387098
Title: NANT Pancreatic Cancer Vaccine: Molecularly Informed Integrated Immunotherapy Combining Innate High-affinity Natural Killer (haNK) Cell Therapy With Adenoviral and Yeast-based Vaccines to Induce T-cell Responses in Subjects With Pancreatic Cancer Who Have Progressed on or After Standard-of-care Therapy
Brief Title: QUILT-3.070:Pancreatic Cancer Vaccine: Subjects With Pancreatic Cancer Who Have Progressed on or After Standard-of-care Therapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-3.070
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Results first posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — ALT-803; avelumab; Bevacizumab; Capecitabine; Cyclophosphamide; Fluorouracil; Leucovorin; 130-nm albumin-bound paclitaxel; Omacor; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NANT Pancreatic Cancer Vaccine (Experimental): A combination of agents will be administered to subjects in this study: Aldoxorubicin HCl, ALT-803, ETBX-011, GI-4000, haNK, avelumab, bevacizumab, capecitabine, cyclophosphamide, fluorouracil, leucovorin, nab-paclitaxel, omega-3-acid ehtyl esters, oxaliplatin, SBRT.
  Interventions: Drug: Aldoxorubicin HCl; Biological: ALT-803; Biological: ETBX-011; Biological: GI-4000; Biological: haNK for infusion; Biological: avelumab; Biological: bevacizumab; Drug: Capecitabine; Drug: Cyclophosphamide; Drug: Fluorouracil; Drug: Leucovorin; Drug: nab-Paclitaxel; Drug: lovaza; Drug: Oxaliplatin; Procedure: SBRT

INTERVENTIONS:
Drug: Aldoxorubicin HCl — Aldoxorubicin hydrochloride
Biological: ALT-803 — Recombinant human super agonist interleukin-15 (IL-15) complex
Biological: ETBX-011 — Ad5 [E1-, E2b-]-CEA
Biological: GI-4000 — Vaccine derived from recombinant Saccharomyces cerevisiae yeast expressing mutant Ras proteins
Biological: haNK for infusion — NK-92 [CD16.158V, ER IL-2]
Biological: avelumab — Recombinant human anti-PD-L1 IgG1 monoclonal antibody
Biological: bevacizumab — Recombinant human anti-VEGF IgG1 monoclonal
Drug: Capecitabine — 5'-deoxy-5-fluoro-N-[(pentyloxy) carbonyl]-cytidine
Drug: Cyclophosphamide — 2-[bis(2-chloroethyl)amino]tetrahydro-2H-1,3,2-oxazaphosphorine 2-oxide monohydrate
Drug: Fluorouracil — 5-fluoro-2,4 (1H,3H)-pyrimidinedione
Drug: Leucovorin — L-Glutamic acid, N-[4-[[(2-amino-5-formyl-1,4,5,6,7,8-hexahydro-4-oxo-6-pteridinyl)methyl]amino]benzoyl]-, calcium salt
Drug: nab-Paclitaxel — Benzenepropanoic acid, β-(benzoylamino)-α-hydroxy-(2aR, 4S, 4aS, 6R, 9S, 11S, 12S, 12aR, 12bS)-6,12b-bis(acetyloxy)-12-(benzoyloxy)-2a, 3, 4, 4a, 5, 6, 9, 10, 11, 12, 12a, 12b-dodecahydro-4,11-dihydroxy-4a, 8, 13, 13-tetramethyl-5-oxo-7,11-methano-1H-cyclodeca[3,4]benz[1,2-b]oxet-9-y1ester,(αR,βS)-(9CI) bound to albumin
Drug: lovaza — Omega-3-acid ethyl esters
Drug: Oxaliplatin — cis-[(1 R,2 R)-1,2-cyclohexanediamine-N,N'] [oxalato(2-)- O,O'] platinum
Procedure: SBRT — Stereotactic Body Radiation Therapy

SUMMARY:
This is a phase 1b/2 study to evaluate the safety and efficacy of metronomic combination therapy in subjects with pancreatic cancer who have progressed on or after previous SoC chemotherapy.

DETAILED DESCRIPTION:
Treatment will be administered in two phases, an induction and a maintenance phase, as described below. Subjects will continue induction treatment for up to 1 year. Treatment in the study will be discontinued if the subject experiences progressive disease (PD) or unacceptable toxicity (not corrected with dose reduction), withdraws consent, or if the Investigator feels it is no longer in the subject's best interest to continue treatment. Those who have a complete response (CR) in the induction phase will enter the maintenance phase of the study. Subjects who experience ongoing stable disease (SD) or an ongoing partial response (PR) at 1 year may enter the maintenance phase at the Investigator's discretion. Subjects may remain on the maintenance phase of the study for up to 1 year. Treatment will continue in the maintenance phase until the subject experiences PD or unacceptable toxicity (not corrected with dose reduction), withdraws consent, or if the Investigator feels it is no longer in the subject's best interest to continue treatment. The maximum time on study treatment, including both the induction and maintenance phases, is 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Able to understand and provide a signed informed consent that fulfills the relevant IRB or Independent Ethics Committee (IEC) guidelines.
3. Histologically-confirmed pancreatic adenocarcinoma with progression on or after SoC therapy.
4. ECOG performance status of 0 to 2.
5. Have at least 1 measurable lesion of ≥ 1.5 cm.
6. Must have a recent formalin-fixed, paraffin-embedded (FFPE) tumor biopsy specimen following the conclusion of the most recent anticancer treatment. If an historic specimen is not available, the subject must be willing to undergo a biopsy during the screening period, if considered safe by the Investigator. If safety concerns preclude collection of a biopsy during the screening period, a tumor biopsy specimen collected prior to the conclusion of the most recent anticancer treatment may be used.
7. Must be willing to provide blood samples prior to the start of treatment on this study.
8. Must be willing to provide a tumor biopsy specimen 8 weeks after the start of treatment, if considered safe by the Investigator.
9. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
10. Agreement to practice effective contraception for female subjects of child-bearing potential and non-sterile males. Female subjects of child-bearing potential must agree to use effective contraception for up to 1 year after completion of therapy, and non-sterile male subjects must agree to use a condom for up to 4 months after treatment. Effective contraception includes surgical sterilization (eg, vasectomy, tubal ligation), two forms of barrier methods (eg, condom, diaphragm) used with spermicide, intrauterine devices (IUDs), and abstinence.

Exclusion Criteria:

1. Serious uncontrolled concomitant disease that would contraindicate the use of the investigational drug used in this study or that would put the subject at high risk for treatment-related complications.
2. Systemic autoimmune disease (eg, lupus erythematosus, rheumatoid arthritis, Addison's disease, autoimmune disease associated with lymphoma).
3. History of organ transplant requiring immunosuppression.
4. History of or active inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis).
5. Inadequate organ function, evidenced by the following laboratory results:

   1. Absolute neutrophil count < 1,000 cells/mm3.
   2. Platelet count < 75,000 cells/mm3.
   3. Total bilirubin greater than the upper limit of normal (ULN; unless the subject has documented Gilbert's syndrome).
   4. Aspartate aminotransferase (AST [SGOT]) or alanine aminotransferase (ALT [SGPT]) > 2.5 × ULN (> 5 × ULN in subjects with liver metastases).
   5. Alkaline phosphatase levels > 2.5 × ULN (> 5 × ULN in subjects with liver metastases, or >10 × ULN in subjects with bone metastases).
   6. Serum creatinine > 2.0 mg/dL or 177 μmol/L.
   7. Serum anion gap > 16 mEq/L or arterial blood with pH < 7.3.
   8. Medically uncorrectable grade 3 anemia (hemoglobin < 8 g/dL).
6. Uncontrolled hypertension (systolic > 160 mm Hg and/or diastolic > 110 mm Hg) or clinically significant (ie, active) cardiovascular disease, cerebrovascular accident/stroke, or myocardial infarction within 6 months prior to first study medication; unstable angina; congestive heart failure of New York Heart Association grade 2 or higher; or serious cardiac arrhythmia requiring medication. Subjects with uncontrolled hypertension should be medically managed on a stable regimen to control hypertension prior to study entry.
7. Serious myocardial dysfunction defined by ECHO as absolute left ventricular ejection fraction (LVEF) 10% below the institution's lower limit of predicted normal.
8. Dyspnea at rest due to complications of advanced malignancy or other disease requiring continuous oxygen therapy.
9. Positive results of screening test for human immunodeficiency virus (HIV).
10. Current chronic daily treatment (continuous for > 3 months) with systemic corticosteroids (dose equivalent to or greater than 10 mg/day methylprednisolone), excluding inhaled steroids. Short-term steroid use to prevent IV contrast allergic reaction or anaphylaxis in subjects who have known contrast allergies is allowed.
11. Known hypersensitivity to any component of the study medication(s).
12. Subjects taking any medication(s) (herbal or prescribed) known to have an adverse drug reaction with any of the study medications.
13. Concurrent or prior use of a strong cytochrome P450 (CYP)3A4 inhibitor (including ketoconazole, itraconazole, posaconazole, clarithromycin, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole, and grapefruit products) or strong CYP3A4 inducers (including phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, and St John's Wort) within 14 days before study day 1.
14. Concurrent or prior use of a strong CYP2C8 inhibitor (gemfibrozil) or moderate CYP2C8 inducer (rifampin) within 14 days before study day 1.
15. Participation in an investigational drug study or history of receiving any investigational treatment within 14 days prior to initiation of treatment on this study, except for testosterone-lowering therapy in men with prostate cancer.
16. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.
17. Concurrent participation in any interventional clinical trial.
18. Pregnant and nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-12-28 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2019-01-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Chan Soon-Shiong Institute for Medicine, El Segundo, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only the Phase 1b portion of the study enrolled participants. The study was terminated early, so no participants were enrolled on the Phase 2 portion of the study.
Groups:
- NANT Pancreatic Cancer Vaccine: The following drugs will be given to the trial participants: GI-4000, haNK, ALT-803, ETBX-011, capecitabine, cyclophosphamide, fluorouracil, leucovorin, nab-paclitaxel, omega-3-acid ethyl esters, oxaliplatin, and SBRT.
  Aldoxorubicin hydrochloride ALT-803: Recombinant human super agonist interleukin-15 (IL-15) complex ETBX-011: Ad5 [E1-, E2b-]-CEA GI-4000: Vaccine derived from recombinant Saccharomyces cerevisiae yeast expressing mutant Ras proteins haNK for infusion: NK-92 [CD16.158V, ER IL-2] avelumab: Recombinant human anti-PD-L1 IgG1 monoclonal antibody bevacizumab: Recombinant human anti-VEGF IgG1 monoclonal Capecitabine: 5'-deoxy-5-fluoro-N-[(pentyloxy) carbonyl]-cytidine
  Cyclophosphamide: 2-[bis(2-chloroethyl)amino]tetrahydro-2H-1,3,2-oxazaphosphorine 2-oxide monohydrate
  Fluorouracil: 5-fluoro-2,4 (1H,3H)-pyrimidinedione
  Leucovorin: L-Glutamic acid, N-[4-[[(2-amino-5-formyl-1,4,5,6,7,8-hexahydro-4-oxo-6-pteridinyl)methyl]amino]benzoyl]-, calcium salt
  nab-Paclitaxel: Benzenepropanoic acid, β-(benzoylamino)-α-hydroxy-(2aR, 4S, 4aS, 6R, 9S, 11S, 12S, 12aR, 12bS)-6,12b-bis(acetyloxy)-12-(benzoyloxy)-2a, 3, 4, 4a, 5, 6, 9, 10, 11, 12, 12a, 12b-dodecahydro-4,11-dihydroxy-4a, 8, 13, 13-tetramethyl-5-oxo-7,11-methano-1H-cyclodeca[3,4]benz[1,2-b]oxet-9-y1ester,(αR,βS)-(9CI) bound to albumin
  lovaza: Omega-3-acid ethyl esters
  Oxaliplatin: cis-[(1 R,2 R)-1,2-cyclohexanediamine-N,N'] [oxalato(2-)- O,O'] platinum
  SBRT: Stereotactic Body Radiation Therapy
Period: Overall Study
Arm/Group | NANT Pancreatic Cancer Vaccine
Started | 4
Completed | 0
Not Completed | 4
Not completed — progressive disease | 1
Not completed — Withdrawal by Subject | 2
Not completed — study terminated by sponsor | 1

BASELINE CHARACTERISTICS:
Arm/Group | NANT Pancreatic Cancer Vaccine
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (11.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 2
subjects with pancreatic cancer who have progressed on or after standard-of-care therapy [Count of Participants; unit: Participants] | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs) and Serious AEs (SAEs), Graded Using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03.
Description: Phase 1b primary endpoint
Time Frame: 30 days after last dose, up to 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | NANT Pancreatic Cancer Vaccine
Number analyzed (Participants) | 4
Participants | 4

ADVERSE EVENTS:
Time Frame: Up to 8 months (30 days after the subject's last dose of study treatment)
Arm/Group | NANT Pancreatic Cancer Vaccine
All-Cause Mortality (participants affected / at risk) | 2/4
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NANT Pancreatic Cancer Vaccine (N=4)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Gastric fistula (Gastrointestinal disorders) | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NANT Pancreatic Cancer Vaccine (N=4)
Fatigue (General disorders) | 4
Injection site reaction (General disorders) | 4
chills (General disorders) | 3
Mucosal inflamation (General disorders) | 3
Pyrexia (General disorders) | 3
Asthenia (General disorders) | 2
Influenza like illness (General disorders) | 1
Injection Site Pain (General disorders) | 1
Odema peripheral (General disorders) | 1
Pain (General disorders) | 1
weight decreased (Investigations) | 3
Eosinophil count increased (Investigations) | 1
Neutophil count decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to low enrollment. Only the safety data is provided.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/98/NCT03387098/Prot_SAP_000.pdf